CLINICAL TRIAL: NCT02338531
Title: Biomarker Research Study for PF-03084014 in cHEmoresistant Triple-negative Breast cAncer
Acronym: RHEA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the discontinuation of the development of the Notch inhibitor PF-03084014-04
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-TNBC-1-RHEA; 2014-004358-32 (EudraCT Number)
Record Dates: First submitted 2015-01-05; First posted 2015-01-14 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapeutic regimen (Experimental): oral administration of PF-03084014, 9 days at 150 mg q.d. (day 1 and 9) and 150 b.i.d. (day 2 till 8)
  Interventions: Drug: PF-03084014; Procedure: Breast cancer surgery

INTERVENTIONS:
Drug: PF-03084014
Procedure: Breast cancer surgery

SUMMARY:
This is a phase II open label Biomarker Research Study off PF-03084014 in non-metastatic triple-negative breast cancer patients with residual disease (cHEmoresistant) after completion of standard neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Female.
3. Histological diagnosis of triple-negative breast cancer (TNBC) breast adenocarcinoma (ER<1%, PR<1% by (IHC) and HER-2 0-1+ by IHC or IHC 2+ and FISH or CISH negative per updated ASCO guidelines).
4. No clinical or radiologic evidence of distant metastasis.
5. Presence of residual primary disease of at least 1.5 cm by U/S or MRI within 14 days preceding the last cycle of standard anthracycline and taxane-based neoadjuvant chemotherapy.

   Patients with synchronous synchronous bilateral cancer and unilateral multifocal or multicentric or bilateral disease breast cancer will be allowed provided histologic diagnosis of TNBC is found on all performed biopsies.
6. Completion of standard anthracycline and taxane-based neoadjuvant chemotherapy. The use of platinum agents in combination with standard neoadjuvant chemotherapy is allowed.
7. ECOG Performance Status (PS) 0 or 1
8. Adequate Bone Marrow Function: Absolute Neutrophil Count (ANC) ≥ 1500/μL or ≥1.5 x 109/L; Platelets ≥100000/μL or ≥100 x 109/L; Hemoglobin ≥ 9 g/dL.
9. Adequate Renal Function: Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥ 60 ml/min.
10. Adequate Liver Function:Total serum bilirubin ≤ 1.0 x ULN or ≤ 2 x ULN in cases of known Gilberts syndrome; Aspartate and Alanine Aminotransferase (AST and ALT) ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN.
11. For patients of childbearing potential: negative serum/urine pregnancy test and use accepted forms of non-hormonal contraception during the study period and up to 6 months after treatment completion.

Exclusion Criteria:

1. Concurrent anti-cancer therapy for current breast cancer (hormone therapy, chemotherapy, radiotherapy, immunotherapy). Patients already included in another therapeutic trial involving an experimental drug.
2. Pregnant or lactating women.
3. Any prior history of invasive breast cancer.
4. Any previous history of non-breast malignancies (excepted basal cell carcinoma or squamous cell carcinoma of the skin) in the preceding 5 years.
5. Known hypersensitivity to the study drug or excipients.
6. Patients with other concurrent severe and/or uncontrolled medical disease or infection which could compromise participation in the study.
7. Subjects unable to swallow oral medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
HES4 gene expression level | tumour tissue samples before study drug and after 9 days of study drug. General analysis after all patients included.
  To demonstrate that PF-03084014 is able to modulate the Notch pathway by down-regulating the expression of the tumor HES4 gene in chemoresistant TNBC (evaluable population).

SECONDARY OUTCOMES:
Safety: General assesment of number and grade of adverse events after short(9-day) administration of oral PF-03084014 in patients with chemoresistant TNBC. | adverse events followed up to 28 days after last PF-03084014 dose.
  Patients will be followed for Adverse Events and Serious Adverse Events from the first dose of study drug up to 28 days after the last dose.
Transcriptome analysis (changes in the HES4 gene expression and tumor transcriptome) | tissue samples before study drug and after 9 days of study drug. General analysis after all patients included.
  To assess changes in the HES4 gene expression and tumor transcriptome for all patients registered in the RHEA study (intent-to-treat population)

CONTACTS AND LOCATIONS:
Overall Officials: Michail Ignatiadis, MD, PhD, Study Director — Medical Oncology Department
Locations (5):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - CMSE, Namur
- France (2):
  - Institut Curie, Paris
  - Institut de Cancérologie Gustave Roussy, Villejuif